CLINICAL TRIAL: NCT05524597
Title: Writing About Experiences and Health in Older Adults II
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Naomi Eisenberger, Professor of Psychology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R01AG071498 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Social Psychology

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Writing about Experiences (Experimental): Participants will be asked to write about experiences with familiar individuals in their lives.
  Interventions: Behavioral: Writing Intervention
- Writing about Places (Placebo Comparator): Participants will be asked to write about experiences with familiar places in their lives.
  Interventions: Behavioral: Writing Intervention

INTERVENTIONS:
Behavioral: Writing Intervention — Participants will be asked to write about different kinds of experiences.

SUMMARY:
UCLA researchers looking for healthy older adults (aged 65+) to participate in a study investigating how writing about experiences can affect your brain and body.

Once a week for 6 weeks, participants will write about their experiences and fill out online questionnaires. Participants will also come to the UCLA campus to complete a neuroimaging session (fMRI), provide a blood spot sample, and fill out questionnaires 2 times: once prior to the 6-week writing period and once immediately after the 6-week writing period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age 65 years and older

Exclusion Criteria:

1. current smokers
2. active, uncontrolled medical disorders
3. chronic infection (e.g., Hepatitis C, HIV)
4. use of certain medications (steroid use, opioid use)
5. psychiatric disorders (e.g., current major depression, bipolar disorder)
6. body mass index (BMI) greater than 35
7. left-handed
8. claustrophobic
9. metal in body

Other exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Distress | Baseline, 6 weeks, 10 weeks
  Composite measure of depression, anxiety, stress (Beck Depression Inventory, Spielberger Trait Anxiety, and Perceived Stress Scale)
Change in Social Support | Baseline, 6 weeks, 10 weeks
  measure of perceived social support (Social Provisions Scale)
Change in Social Participation | Baseline, 6 weeks, 10 weeks
  measure of participation in social activities (Lifestyle Activities Questionnaire)
Change in Inflammatory Gene Expression | Baseline, 6 weeks, 10 weeks
  changes in proinflammatory gene expression
Change in Dorsal Anterior Cingulate Cortex (dACC) Activity in response to stress | Baseline, 6 weeks
  Parameter estimates from dACC region-of-interest
Change in Anterior Insula Activity in response to stress | Baseline, 6 weeks
  Parameter estimates from bilateral anterior insula region-of-interest
Change in Amygdala Activity in response to threat | Baseline, 6 weeks
  Parameter estimates from bilateral amygdala region-of-interest
Change in Ventral Striatum Activity in response to prosocial behavior | Baseline, 6 weeks
  Parameter estimates from bilateral ventral striatum region-of-interest
Change in Septal Area Activity in response to prosocial behavior | Baseline, 6 weeks
  Parameter estimates from septal area region-of-interest

SECONDARY OUTCOMES:
Change in Memory | Baseline, 6 weeks, 10 weeks
  changes in recall ability (Montreal Cognitive Assessment Test)
Change in Beliefs about Aging | Baseline, 6 weeks, 10 weeks
  changes in cognitive, affective, and social beliefs about aging (Expectations Regarding Aging survey)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cognitive Neuroscience, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No